CLINICAL TRIAL: NCT03478566
Title: The Diagnostic Accuracy and Reliability of Transcutaneous Carbon Dioxide Monitoring at Home for Nocturnal Hypoventilation Screening in Children With Neuromuscular Disease
Brief Title: Transcutaneous CO2 Monitoring at Home for Children With Neuromuscular Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Staff Physician, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000059242
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Sleep Disorder; Breathing-Related; Central Apnea; Neuromuscular Diseases; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea, Central; Neuromuscular Diseases; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcutaneous CO2 monitoring (Experimental)
  Interventions: Device: Transcutaneous CO2 monitoring

INTERVENTIONS:
Device: Transcutaneous CO2 monitoring — The aim is to assess the accuracy of ambulatory, at home, transcutaneous CO2 monitoring in pediatric Neuromuscular Disease (NMD).

SUMMARY:
There is an unmet demand for the evaluation of nocturnal hypoventilation in children with NMD. An ambulatory screening tool that can reliably facilitate timely diagnosis and treatment in these children would be invaluable. If an ambulatory, at home, tcCO2 monitoring device is shown to be diagnostically accurate, sleep physicians would be able to triage children on existing waiting lists and optimize screening of nocturnal hypoventilation as recommended by international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* children with a confirmed diagnosis of NMD that meet criteria for evaluating SDB as per international recommendations
* lives within the greater Toronto area.

Exclusion Criteria:

* known diagnosis of nocturnal hypoventilation
* current ventilatory support
* physician diagnosis of active upper respiratory tract infection (fever, increased cough, rhinorrhea, increased nasal congestion, sore throat, headache, malaise and/or sneezing).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of ambulatory, at home, transcutaneous CO2 (tcCO2) monitoring to diagnose nocturnal hypoventilation as compared to the gold standard, end tidal CO2 conducted during polysomnogram (PSG). | 9 months

SECONDARY OUTCOMES:
a) Agreement of tcCO2 monitoring when worn in the ambulatory, at home, setting compared to tcCO2 recorded during a PSG in a hospital based sleep laboratory for diagnosis of nocturnal hypoventilation. | 9 months
  b) Correlation of the pre and post sleep capillary blood gas results with end tidal CO2 (etCO2) and tcCO2 recordings during PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, Principal Investigator — Staff Physician
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi J, Chiang J, Ambreen M, Snow N, Mocanu C, McAdam L, Goldstein RS, Rose L, Amin R. Ambulatory transcutaneous carbon dioxide monitoring for children with neuromuscular disease. Sleep Med. 2023 Jan;101:221-227. doi: 10.1016/j.sleep.2022.10.028. Epub 2022 Nov 2. PMID 36435158